CLINICAL TRIAL: NCT04545294
Title: Online Left-hemispheric Frontoparietal Theta In-phase tACS During Working Memory Training in Schizophrenia Patients: A Pilot Randomized Double-blind, Sham-controlled Study of the Effects on Negative Symptoms
Brief Title: Theta tACS During Working Memory Training: A Pilot Study of the Effects on Negative Symptoms of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-An Chang, MD, Attending Psychiatrist, Department of Psychiatry, Principal Investigator, Associate Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2-106-05-123
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Negative Symptoms; Working Memory Training; Psychosocial Impairment; Autonomic Imbalance; EEG
Keywords: Schizophrenia; Schizoaffective Disorder; Transcranial alternating current stimulation; Theta oscillatory rhythm; Theta Phase-Coupling; Negative symptoms; Working memory training
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation concealment was further ensured by the administration of tACS using "study mode of the device" in which a five-digit numerical code specific to individual participant was entered into the device (Eldith DC stimulator Plus, NeuroConn, Ilmenau, Germany) that resulted in either active or sham stimulation, i.e., the researcher got the randomization code and a unique five-digit numerical code for an individual participant from the study coordinator while tACS administrator entered the code for study mode into the device. The study coordinator had continuous access to the randomization list and unblinded the study after the final visit of the last participant. Not until the unblinding of the trial did the participants, tACS administrators, researchers and clinical raters know the actual stimulation types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active theta (6Hz) in-phase tACS (Experimental): θ tACS will be administered during the dual n-back task, starting at the beginning of each task and lasting for 20 min. In the active θ tACS condition, sinusoidal tACS will be delivered by two battery-operated devices (Eldith DC stimulator Plus, neuroConn, Ilmenau, Germany) connected with two 4 × 1 wire adaptors (Equalizer Box, NeuroConn, Ilmenau, Germany), via 10 carbon rubber electrodes (1 cm radius, high-definition 4 × 1 rings configuration with a gel layer of 2.0 mm), at 6 Hz frequency, 2 mA current intensity without DC offset, with 100 cycles ramp-up/ramp-down and a 0° relative phase, for 20 min, twice-daily on 5 consecutive weekdays.
  Interventions: Device: Theta tACS
- Sham tACS (Sham Comparator): During sham sessions, tACS will be applied in the synchronous condition for 30 s of 2 mA normal-like stimulation at the beginning of each dual n-back task. After that, only a tiny current pulse (110 μA over 15 ms) for impedance control took place every 550 ms during the remaining time.
  Interventions: Device: Theta tACS

INTERVENTIONS:
Device: Theta tACS — See detail in arm/group descriptions regarding the intervention.

SUMMARY:
In this randomized double-blind trial, we investigated whether externally induced left-hemispheric frontoparietal theta synchronization by multi-electrode online theta (6Hz) transcranial alternating current stimulation (tACS) would enhance the influence of a working memory training on negative symptoms of schizophrenia.

DETAILED DESCRIPTION:
Negative symptoms have a negative impact on the prognosis of schizophrenia, but effective treatment for this symptom dimension is still under investigation. Identifying a treatment target that has a close link to negative symptoms or highly impacts negative symptoms may help to develop an effective therapy to counteract negative symptoms of schizophrenia. Recent theoretical and empirical work linking negative symptoms and cognitive impairment in schizophrenia has identified a potential treatment target: cognitive deficits. Evidence has indicated that cognitive remediation (CR) has a positive effect on improving negative symptoms of schizophrenia, in particular behavioural negative symptoms.

Although it is still debated which active components of CR contribute to the improvements in negative symptoms. The framework proposed by Gold and colleagues may be a candidate to explain how CR improves negative symptoms (i.e., possible through improving working memory). Anhedonia (i.e., the diminished ability to experience pleasure and reduced reactivity to pleasurable stimuli) represents a challenging negative symptom in schizophrenia.The impairment in hedonic processing has been associated with reduced motivation to engage in potentially rewarding events. Working memory (WM) plays an important role in the formation, maintenance, and retrieval of affective and value representations, all of which are essential for anticipatory pleasure. Individuals represent events and forecast pleasure by using WM in order to recruit motivational resources. It has been suggested that there is a hedonic detector system within the WM model and that WM serves as a potential underlying cognitive mechanism for anticipatory pleasure and goal-related behaviours. Problems in WM may reduce the ability to retrieve and manipulate information to motivate and guide future behaviour, thereby contributing to diminished motivation and the pleasure experience. It is known that the recruitment of the prefrontal-striatal system (including dorsolateral prefrontal cortex, cingulate cortex, insula, and ventral striatum) implicates in hedonic processing. It is also known that the same brain regions can be viewed as core brain regions of the WM network because they are activated during WM load. The overlap in activation of the prefrontal-striatal system during hedonic processing and WM provides robust evidence supporting the relationship between hedonic capacity and WM. Evidence indicated a correlation between the activity in WM brain networks and the improvement in negative symptoms following antipsychotic treatment, suggesting a mediating effect of WM on negative symptoms improvement in the context of a pharmacological intervention. More recently, studies indicated that 20 sessions of WM training (dual n-back task training) showed neural transfer effect to enhance hedonic processing in individuals with high social anhedonia and ameliorate hedonic dysfunction in schizophrenia patients with prominent negative symptoms.

In addition to WM training, non-invasive brain stimulation (NIBS) is also a non-pharmacological method to improve brain neural plasticity. For example, repetitive transcranial magnetic stimulation (rTMS) can change the activity of cortical nerve temporarily or continuously and enhance neural plasticity. However, the ability of rTMS alone to improve cognitive function in schizophrenia is frequently limited to some extent, necessitating a combination with WM training to boost cognitive functions.

Transcranial alternating current stimulation (tACS), a safe NIBS technique that applies low-intensity alternating current, is also a potential therapeutic option in treating the cognitive impairment in schizophrenia. The stimulation frequency of tACS is usually set to coincide with the targeted brain endogenous rhythms. It would synchronize the neural oscillations in the stimulated cortical regions to the applied stimulation frequency. Different tACS current intensity (0.5 to 4 mA), stimulation frequency (0.1 to 80 Hz), electrode montages, phase difference across the stimulation site, with/without DC offset, and the states (e.g., at rest or concurrently under the tasks) during stimulation contribute to its different effects. If both the target electrode and the reference electrode are in the same phase of the cycle of the current at any given time, the phase difference will be 0 degree (i.e., in-phase). The phase difference will be 180 degrees (i.e., anti-phase) if the electrodes are in the opposite phase. In-phase and anti-phase tACS over brain regions elicits synchronization and desynchronization of neuronal activity across the brain regions, respectively.

The state-dependent tACS effects indicate that the effects of tACS are enhanced when the state of the targeted brain regions is active. Specifically, synchronization of frontoparietal regions at theta frequencies dominates during an executive task. tACS at the frequency close to the theta oscillation activated by an executive task would elicit more resonance and may, in turn, help to enhance executive function. tACS applied when an individual is concurrently engaged in a specific cognitive task is defined as online tACS. In healthy subjects, online theta (6Hz) in-phase tACS facilitated frontoparietal phase coupling (synchronization) resulting in improved WM performance, whereas online theta (6Hz) anti-phase tACS disrupted theta phase-coupling (desynchonization) resulting in impaired WM performance.

The prolonged after-effects of tACS may be related to a phenomenon called spike-timing-dependent plasticity (STDP), a process that modifies the connection strengths based on the relative timing of the input and output spikes (or action potentials) of a neuron. STDP means that synapse will be strengthened if input action potentials occur immediately before the output action potentials, and synapse will be made weaker if an input action potentials occur immediately after an output action potentials. The STDP process is known to explain in part long-term depression (LTD) and long-term potentiation (LTP) of nervous systems. To sum up, tACS at a frequency close to that of resonance frequency during tACS may intensify the synapses across the stimulated regions through the mechanism of STDP. Repetitive (multiple-session) tACS during specific time intervals may consolidate the neuroplasticity effects, and may, in turn, elicit a long-lasting effect for further clinical application in treating neuropsychiatric disorders. In schizophrenia patients, a few case reports indicated 1-5 sessions of online theta in-phase tACS over left frontoparietal regions improved the performance of WM and several other cognitive domains.

So far, there is no relevant research report exploring whether and how the joint intervention (i.e., online theta (6Hz) in-phase tACS over the left frontoparietal regions plus WM training) will have a combined effect on improving the performance of WM and other cognitive domains in schizophrenic patients. Neither is any research investigating whether online theta (6Hz) in-phase tACS over the left frontoparietal regions can potentiate the effects of WM training on improving negative symptoms of schizophrenia. To sum up, we hypothesize that the combination training mode of active online theta tACS plus WM training would have a greater ability to reduce negative symptoms of schizophrenia compared to the training mode of sham online theta tACS plus WM training. The study aims to test the efficacy of "active online theta tACS plus WM" versus "sham online theta tACS plus WM training" in improving negative symptoms, WM performance, and other cognitive domains performance of schizophrenia using a double-blinded, randomized sham-controlled trial design. In order to evaluate the efficacy of the interventions, we will use behavioral outcomes (e.g., negative symptoms assessment and neurocognitive assessment) and neurophysiological outcomes (e.g., EEG and heart rate variability).

Methods

Dual N back training

The study will use a dual n-back task for WM training. In this task, squares at 8 different locations will show up sequentially (stimulus length, 500 ms; inter-stimulus interval, 2,500 ms) on a computer screen every 3 seconds. Simultaneously with the presentation of the squares, one of eight consonants will show up sequentially through a speaker. Participants will have to judge whether the location of a square and the consonant they heard matches the one n-back before (the same n value for both visual and auditory targets). Each training session has 20 blocks consisting of 20 + n trials and takes around 25 min. Each block includes six auditory and six visual targets (four appearing in only one modality, and two appearing in both modalities simultaneously) whose locations are random. Participants will have to make responses manually by pressing the mouse left-click button for visual targets and the right-click button for auditory targets. No responses were required for non-targets. If a target is correctly detected, a green flash will be given, which constitutes a positive feedback. If a target is falsely detected, a blue flash will be given, which constitutes a negative feedback. The dual N back training is designed to continuously vary its difficulty by modifying the WM load (i.e., the level of n) and thereby track the participants' performance. Each training session begins at n = 1. Participants' performance will be analyzed after each block and the level of n for the next block will be adapted according to the following principle. The level of n increases by 1 in the next block if the mistakes per modality made by the participant are<3. Conversely, n would decrease by 1 if the mistakes per modality made by the participant are>5. In all other cases, the n is kept unchanged. Participants will come to the laboratory and take part in the WM training sessions twice daily for 5 weekdays (total 10 sessions), with each session lasting for approximately 25 minutes. The time interval between twice-daily sessions will be >3 hours.

Online left-hemispheric frontoparietal theta (6Hz) in-phase tACS

θ tACS will be administered during the dual n-back task, starting at the beginning of each task and lasting for 20 min. In the active θ tACS condition, sinusoidal tACS will be delivered by two battery-operated devices connected with two 4 × 1 wire adaptors (Equalizer Box, NeuroConn, Ilmenau, Germany). The electrode montages used for θ tACS will be positioned at left frontoparietal locations. The stimulation electrodes of the 1st stimulator will be placed at the International 10-10 electrode position F1, F5, AF3, and FC3 (stimulation electrodes) and CPz (return electrode) to cover the left frontal cortex. For the 2nd stimulator, the stimulation electrodes will be placed at P1, P5, CP3, and PO3 (stimulation electrodes) and FCz (return electrode) to cover the left parietal cortex. A NeuroConn digital to analog converter (DAQ) will control the two stimulators and create an in-phase (synchronous) setup (0° relative phase difference between the output signals of the two tACS-stimulators).

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants aged 20-65 with DSM-V-defined schizophrenia or schizoaffective disorder.
2. Duration of illness > 2 years.
3. Being clinically stable and on an adequate therapeutic dose of antipsychotics for at least 8 weeks prior to enrolment.
4. Agreement to participate in the study and provide the written informed consent.

Exclusion Criteria:

1. Having unstable medical conditions, current psychiatric comorbidity or active substance use disorder (in exception to caffeine and/or tobacco).
2. Having a history of seizures, meningitis or encephalitis.
3. Having contraindications for transcranial electrical stimulation or transcranial magnetic stimulation, e.g., pacemakers, metallic or magnetic pieces in the head/brain, ear implants and other implantible brain medical devices.
4. Having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases.
5. Pregnancy or breastfeeding at enrollment.
6. Skin lesions on scalp at the area of electrode application

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
The change over time in the negative symptoms subscale score of the Chinese version of the Positive and Negative Syndrome Scale (PANSS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  A clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder. The patient is rated from 1 to 7 on 30 different symptom items. All items scores are summed up to yield a total PANSS score, which ranges from 30 to 210. A higher score indicates greater psychopathological symptom severity. There are 7 items for positive symptoms subscale (score 7-49), 7 items for negative symptoms subscale (score 7-49), 16 items for general symptoms subscale (score 16-112).

SECONDARY OUTCOMES:
The change over time in the Chinese version of the Positive and Negative Syndrome Scale Factor Score for Negative Symptoms (PANSS-FSNS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  A clinician-administered rating scale to measure the severity of psychopathological symptoms of the patients with schizophrenia spectrum disorder. The patient is rated from 1 to 7 on 30 different symptom items. All items scores are summed up to yield a total PANSS score, which ranges from 30 to 210. A higher score indicates greater psychopathological symptom severity. The five-factor PANSS model can be obtained by calculating from 26 of 30 items of PANSS: positive (5 items, P1+P3+P5+P6+G9,score 5-35) , negative (7 items, N1+N2+N3+N4+N6+G7+G16, score 7-49), grandiosity/excitement (4 items, score 4-28), disorganization (5 items, score 5-35), and depression (4 items, score 4-28) factor scores. The cognitive component of the PANSS can be obtained as well (3 items, P2+N5+G11, score 3-21).
The change over time in the score of the Chinese version of the Scale for the Assessment of Negative Symptoms (SANS) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  The Scale for the Assessment of Negative Symptoms (SANS) is used to assess negative symptoms in schizophrenia on a 25 item, 6-point scale. The SANS measures five domains of the negative symptoms including affective flattening or blunting, alogia, avolition - apathy, anhedonia - Asociality, Attention. In each domain, separate symptoms are rated from 0 (absent) to 5 (severe). A total SANS score ranges from 0 to 125.
The change over time in the score of the Chinese version of the Personal and Social Performance scale (PSP) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  A clinician-administered rating scale to measure the psychosocial functioning of the patients with schizophrenia spectrum disorder. The PSP scale measures psychosocial functioning within four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior.The patient is rated from 1 to 6 on each item of the four domains. A higher score indicates greater psychosocial functioning in any of the four domains. The final global score is defined according to a summary instruction table. This scale provides a single, overall rating from 1 to 100, where a higher score represents better personal and social function.
The change over time in the score of the self-reported version of the graphic personal and social performance scale (SRG-PSP) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The SRG-PSP is a self-rating scale of proven validity and reliability, comprising both male and female versions of cartoon-like pictures that are derived from the narrative text of the four domains of Personal and Social Performance (PSP) scale including the sub-items of socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behaviour.
The change over time in the score of the abbreviated version of the Scale to Assess Unawareness in Mental Disorder in schizophrenia (SUMD) (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  An expert-rating scale based on a patient interview to measure patients' clinical insight. The abbreviated version of SUMD comprises 9 items measuring current states of awareness as follows: (1) a mental disorder, (2) consequences of a mental disorder, (3) effects of drugs, (4) hallucinatory experiences, (5) delusional ideas, (6) disorganized thoughts, (7) blunted affect, (8) anhedonia, and (9) lack of sociability. Scores on each item range from 0 to 3. A score of 0 indicates 'not applicable'; 1, 'aware'; 2, 'somewhat aware/unaware' and 3, 'severely unaware.' Based on the 3 dimensions approach of the abbreviated version of SUMD, the scores on the items 1-3, 4-6 and 7-9 were averaged to obtain the dimension score of 'awareness of the disease', 'awareness of positive symptoms', and 'awareness of negative symptoms', respectively. All dimension scores were linearized on a 0-100 scale, with 0 and 100 indicating the lowest and highest level of unawareness, respectively.
The change over time in the score of the Taiwanese version of the Beck Cognitive Insight Scale (BCIS) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  Cognitive insight was measured by the Taiwanese version of the Beck Cognitive Insight Scale (BCIS), a self-reported instrument comprising 15 items.The Taiwanese BCIS is composed of 2 subscales including reflective attitude (9 items) and certain attitude (6 items). We obtained a R-C (reflective attitude minus certain attitude) index of the Taiwanese BCIS, representing the measurement of cognitive insight by subtracting the score of the certain attitude subscale from that of the reflective attitude subscale. Lower R-C index scores indicate poorer cognitive insight.
The change over time in the score of the Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The Taiwanese version of the Self-Appraisal of Illness Questionnaire (SAIQ) was used to assess attitudes toward mental illness and experience of psychiatric treatment.This self-administered tool was composed of 17 items. The patients rated the extent to which they agreed with each statement of the item by using a four-point Likert scale, ranging from 1, ''do not agree at all'', to 4, ''completely agree''. Whether the scale score is in order from least to most or from the most to least depends on the content of the item statement. The total score of SAIQ ranges from 17 to 68.
The change over time in the negative symptoms subscale score of the Chinese version of the Schizophrenia Quality of Life Scale Revision Four (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The Chinese version of the Schizophrenia Quality of Life Scale Revision Four is a self-administered questionnaire of 33 items in two domains: psychosocial and vitality. All but four items are coded on a scale of 0-4 according to the frequency of occurrence during the previous 7 days (0 = always, 4 = never; the four exceptions are coded 0 = never, 4 = always). A higher score indicates higher health-related QoL.
The changes over time in the results of Digit span (forward and backward) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A test to measure the capacity of working memory of the patients
The changes over time in the results of Finger tapping test (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test that examines motor functioning, specifically, motor speed and lateralized coordination.
The changes over time in the results of Continuous Performance (CPT, version 2.0) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test that examines the performance of prefrontal-mediated task
The changes over time in the results of Wisconsin Card Sorting Test (WCST) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement.
The changes over time in the results of Tower of London test (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  A neuropsychological test for the assessment of executive functioning specifically to detect deficits in planning, which may occur due to a variety of medical and neuropsychiatric conditions.
The changes over time in the results of Color Trails Test (CTT) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  The CTT, a culture-neutral version of the Trail Making Test, was selected to measure sustained visual attention. The CTT consists of two parts (CTT-1 and CTT-2). The CTT-1 requires participants to connect a series of numbered circles that are randomly printed on a sheet of paper. In the CTT-2, numbered circles of 1 to 25 are shown twice (printed in pink and in yellow) randomly on a sheet of paper. Participants are asked to connect the numbers from 1 to 25 alternating between the two colors.
The changes over time in the results of Stroop Color Word Test (SCWT) (from baseline to the timepoints immediately after intervention and at one-week follow-up) | Two weeks
  Stroop Color Word Test (SCWT), Chinese version; was administered to measure selective attention and cognitive flexibility. SCWT is composed of three parts, each lasting for 45 seconds.
The changes over time in the results of the dual 2-back task (from baseline to the timepoints immediately after intervention, at one-week and one-month follow-ups). | Five weeks
  In the dual 2-back task, squares at 8 different locations will show up sequentially (stimulus length, 500 ms; inter-stimulus interval, 2,500 ms) on a computer screen every 3 seconds. Simultaneously with the presentation of the squares, one of eight consonants will show up sequentially through a speaker. Participants will have to judge whether the location of a square and the consonant they heard matches the one 2-back before (the same for both visual and auditory targets). Each experimental condition was presented with 100+n trials, resulting in a task time of 5 min. Each task includes 30 auditory and 30 visual targets (four appearing in only one modality, and two appearing in both modalities simultaneously) whose locations are random. Participants will have to make responses manually by pressing the mouse left-click button for visual targets and the right-click button for auditory targets. No responses were required for non-targets.
The changes over time in indices of heart rate variability (HRV) measured at baseline, during the first session of tACS, after 10-session tACS, at 1-week and 1-month follow-ups. | Five weeks
  HRV indices represent autonomic functioning. ECG electrodes were placed on bilateral arms just below the elbows, with a ground electrode placed just above the right wrist bone. Lead I electrocardiogram of each patient was taken for 5 min after sitting and having a rest for 20 min in a soundproof, dim-lighted room with thermostatic control. At the four timepoints (baseline, after 10-session tACS, at 1-week and 1-month follow-ups), HRV will be collected during resting and during a dual 2-back task. The ECG signals were acquired, stored, pre-processed according to the recommended procedures and processed by an HRV analyser (LR8Z11, Yangyin Corp., Taipei, Taiwan). The time domain of HRV is obtained: Standard deviation of NN intervals (SDNN). Power spectrum of HRV is quantified into the standard frequency-domain measurements including low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15-0.40 Hz).
The changes over time in EEG absolute power and coherence in the frontoparietal electrode pairs in the alpha and theta range (from baseline to the timepoints after intervention, at one-week and one-month follow-ups) | Five weeks
  In a recliner in a dimly lit, electrically shielded room, patients' EEGs were recorded at 4 timepoints (baseline, after 10-session tACS, at 1-week and 1-month follow-ups) by using the Neuro Prax® TMS/tDCS full-band DC-EEG system with 32 EEG Ag/AgCl electrodes in the standard 10-20 International placement. EEG will be collected during resting, eye-opened (5min) and during a dual 2-back task (5min). Signals will be amplified in the dynamic input range of ± 140 mV at a resolution of 0.5 μV by using EEG amplifiers and stored for offline analyses. Eye or muscle artifacts were automatically detected and removed using NeuroPrax's built-in software.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Chang, M.D., Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

REFERENCES:
- [Background] Alagapan S, Schmidt SL, Lefebvre J, Hadar E, Shin HW, Frӧhlich F. Modulation of Cortical Oscillations by Low-Frequency Direct Cortical Stimulation Is State-Dependent. PLoS Biol. 2016 Mar 29;14(3):e1002424. doi: 10.1371/journal.pbio.1002424. eCollection 2016 Mar. PMID 27023427
- [Background] Battleday RM, Muller T, Clayton MS, Cohen Kadosh R. Mapping the mechanisms of transcranial alternating current stimulation: a pathway from network effects to cognition. Front Psychiatry. 2014 Nov 20;5:162. doi: 10.3389/fpsyt.2014.00162. eCollection 2014. No abstract available. PMID 25477826
- [Background] Cella M, Preti A, Edwards C, Dow T, Wykes T. Cognitive remediation for negative symptoms of schizophrenia: A network meta-analysis. Clin Psychol Rev. 2017 Mar;52:43-51. doi: 10.1016/j.cpr.2016.11.009. Epub 2016 Nov 28. PMID 27930934
- [Background] Farreny A, Aguado J, Ochoa S, Haro JM, Usall J. The role of negative symptoms in the context of cognitive remediation for schizophrenia. Schizophr Res. 2013 Oct;150(1):58-63. doi: 10.1016/j.schres.2013.08.008. Epub 2013 Aug 29. PMID 23993864
- [Background] Fusar-Poli P, Papanastasiou E, Stahl D, Rocchetti M, Carpenter W, Shergill S, McGuire P. Treatments of Negative Symptoms in Schizophrenia: Meta-Analysis of 168 Randomized Placebo-Controlled Trials. Schizophr Bull. 2015 Jul;41(4):892-9. doi: 10.1093/schbul/sbu170. Epub 2014 Dec 20. PMID 25528757
- [Background] Gold JM, Barch DM, Carter CS, Dakin S, Luck SJ, MacDonald AW 3rd, Ragland JD, Ranganath C, Kovacs I, Silverstein SM, Strauss M. Clinical, functional, and intertask correlations of measures developed by the Cognitive Neuroscience Test Reliability and Clinical Applications for Schizophrenia Consortium. Schizophr Bull. 2012 Jan;38(1):144-52. doi: 10.1093/schbul/sbr142. Epub 2011 Nov 17. PMID 22101961
- [Background] Gold JM, Waltz JA, Prentice KJ, Morris SE, Heerey EA. Reward processing in schizophrenia: a deficit in the representation of value. Schizophr Bull. 2008 Sep;34(5):835-47. doi: 10.1093/schbul/sbn068. Epub 2008 Jun 30. PMID 18591195
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Klimesch W. EEG alpha and theta oscillations reflect cognitive and memory performance: a review and analysis. Brain Res Brain Res Rev. 1999 Apr;29(2-3):169-95. doi: 10.1016/s0165-0173(98)00056-3. PMID 10209231
- [Background] Kringelbach ML, Berridge KC. Towards a functional neuroanatomy of pleasure and happiness. Trends Cogn Sci. 2009 Nov;13(11):479-87. doi: 10.1016/j.tics.2009.08.006. Epub 2009 Sep 24. PMID 19782634
- [Background] Lett TA, Voineskos AN, Kennedy JL, Levine B, Daskalakis ZJ. Treating working memory deficits in schizophrenia: a review of the neurobiology. Biol Psychiatry. 2014 Mar 1;75(5):361-70. doi: 10.1016/j.biopsych.2013.07.026. Epub 2013 Sep 5. PMID 24011822
- [Background] Li X, Chu MY, Lv QY, Hu HX, Li Z, Yi ZH, Wang JH, Zhang JY, Lui SSY, Cheung EFC, Shum DHK, Chan RCK. The remediation effects of working memory training in schizophrenia patients with prominent negative symptoms. Cogn Neuropsychiatry. 2019 Nov;24(6):434-453. doi: 10.1080/13546805.2019.1674644. Epub 2019 Oct 4. PMID 31583951
- [Background] Li X, Li Z, Li K, Zeng YW, Shi HS, Xie WL, Yang ZY, Lui SS, Cheung EF, Leung AW, Chan RC. The neural transfer effect of working memory training to enhance hedonic processing in individuals with social anhedonia. Sci Rep. 2016 Oct 18;6:35481. doi: 10.1038/srep35481. PMID 27752140
- [Background] Li X, Xiao YH, Zou LQ, Li HH, Yang ZY, Shi HS, Lui SS, Cheung EF, Chan RC. The effects of working memory training on enhancing hedonic processing to affective rewards in individuals with high social anhedonia. Psychiatry Res. 2016 Nov 30;245:482-490. doi: 10.1016/j.psychres.2016.09.006. Epub 2016 Sep 8. PMID 27639163
- [Background] Nejad AB, Madsen KH, Ebdrup BH, Siebner HR, Rasmussen H, Aggernaes B, Glenthoj BY, Baare WF. Neural markers of negative symptom outcomes in distributed working memory brain activity of antipsychotic-naive schizophrenia patients. Int J Neuropsychopharmacol. 2013 Jul;16(6):1195-204. doi: 10.1017/S1461145712001253. Epub 2012 Nov 20. PMID 23164479
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259
- [Background] Rottschy C, Langner R, Dogan I, Reetz K, Laird AR, Schulz JB, Fox PT, Eickhoff SB. Modelling neural correlates of working memory: a coordinate-based meta-analysis. Neuroimage. 2012 Mar;60(1):830-46. doi: 10.1016/j.neuroimage.2011.11.050. Epub 2011 Dec 1. PMID 22178808
- [Background] Sreeraj VS, Shanbhag V, Nawani H, Shivakumar V, Damodharan D, Bose A, Narayanaswamy JC, Venkatasubramanian G. Feasibility of Online Neuromodulation Using Transcranial Alternating Current Stimulation in Schizophrenia. Indian J Psychol Med. 2017 Jan-Feb;39(1):92-95. doi: 10.4103/0253-7176.198937. PMID 28250567
- [Background] Sreeraj VS, Shivakumar V, Sowmya S, Bose A, Nawani H, Narayanaswamy JC, Venkatasubramanian G. Online Theta Frequency Transcranial Alternating Current Stimulation for Cognitive Remediation in Schizophrenia: A Case Report and Review of Literature. J ECT. 2019 Jun;35(2):139-143. doi: 10.1097/YCT.0000000000000523. PMID 30024457
- [Background] Strauss GP. Translating basic emotion research into novel psychosocial interventions for anhedonia. Schizophr Bull. 2013 Jul;39(4):737-9. doi: 10.1093/schbul/sbt082. Epub 2013 May 24. No abstract available. PMID 23709387
- [Background] Vinograd M, Craske MG. Using Neuroscience to Augment Behavioral Interventions for Depression. Harv Rev Psychiatry. 2020 Jan/Feb;28(1):14-25. doi: 10.1097/HRP.0000000000000241. PMID 31913979
- [Background] Vossen A, Gross J, Thut G. Alpha Power Increase After Transcranial Alternating Current Stimulation at Alpha Frequency (alpha-tACS) Reflects Plastic Changes Rather Than Entrainment. Brain Stimul. 2015 May-Jun;8(3):499-508. doi: 10.1016/j.brs.2014.12.004. Epub 2014 Dec 20. PMID 25648377
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168